CLINICAL TRIAL: NCT03924401
Title: Acute GVHD Suppression Using Costimulation Blockade to Expand Non-malignant Transplant (ASCENT)
Brief Title: Acute GVHD Suppression Using Costimulation Blockade to Expand Non-malignant Transplant
Acronym: ASCENT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Thrasher Research Fund (Other); Sickle Cell Transplant Advocacy & Research Alliance (STAR) (Unknown); Aflac Cancer and Blood Disorders Center (Unknown); Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, John T. Horan, MD, MPH, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00108549
Record Dates: First submitted 2019-04-19; First posted 2019-04-23 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Graft Versus Host Disease
Keywords: Pediatrics; Non-malignant hematologic diseases; Severe aplastic anemia; Fanconi anemia; Sickle cell disease; Hematopoietic stem cell transplantation; Thalassemia; Mismatched unrelated donor; Matched unrelated donor
MeSH Terms: conditions — Graft vs Host Disease; Anemia, Aplastic; Fanconi Anemia; Anemia, Sickle Cell; Thalassemia | interventions — Abatacept

STUDY DESIGN:
Intervention Model Description: The trial will include two strata: one for patients with a 7/8 matched donor and one for those with a matched 8/8 donor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants Receiving Abatacept (Experimental): Pediatric participants who are undergoing URD HSCT for serious NMHD will receive 8 doses of abatacept in addition to conventional GVHD prophylaxis.
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — All patients will receive 8 doses of abatacept (10 mg/kg intravenously on days -1, +5, +14, +28, +56, +84, +112, and +150) in addition to conventional GVHD prophylaxis.
  Other Names: Orencia

SUMMARY:
This trial will see if extended abatacept administration (combined with a standard regimen of tacrolimus and mycophenolate mofetil) will prevent acute and chronic graft-versus-host disease (GVHD) in children and adolescents receiving unrelated donor (URD) hematopoietic stem cell transplantation (HSCT), without compromising their engraftment or reconstitution of protective immunity to infection.

The study will enroll 30 pediatric patients with serious non-malignant hematologic diseases (NMHD) undergoing URD HSCT. The trial will include patients with 7/8 donors and those with 8/8 (matched) donors. All participants will receive 8 doses of abatacept. Recruitment is expected to last for about 2 years and participants will be followed for up to 3 years.

DETAILED DESCRIPTION:
Many serious non-malignant hematologic diseases (NMHD) affecting children, including severe aplastic anemia (SAA), Fanconi anemia (FA), sickle cell disease (SCD), and thalassemia can be cured by allogeneic hematopoietic stem cell transplantation (HSCT). While the best results are achieved with HSCT from human leukocyte antigen (HLA)-matched siblings, most children lack such donors, and many children with NMHD are therefore transplanted with grafts from an adult unrelated donor (URD). Because URD grafts are less histocompatible, they are more likely to cause GVHD, a process driven by the reaction of donor T cells against incompatible host tissues. Despite the routine administration of immune suppression for GVHD prophylaxis, GVHD claims the lives of many and plagues others with incapacitating chronic illness. For NMHD, the threat of GVHD limits the use of URD HSCT to only the most severely affected children. In African-Americans and other ethnic minorities, the situation is compounded by the fact that most of these children lack fully matched URD and typically receive mismatched and matched grafts, which carry an increased risk for graft rejection. A more effective form of GVHD prophylaxis that does not compromise engraftment is urgently needed, both to improve outcomes for those children undergoing HSCT as well as to allow expansion of this curative therapy to the many children with NMHD who forego transplantation because of the risk for GVHD.

The researchers have investigated the use of the co-stimulation blocking agent CTLA4-Ig (abatacept) to prevent GVHD. Study results to date indicate that abatacept strongly inhibits allo-reactive donor T cells and is clinically safe and effective. The clinical experience has included a variety of recipients: children and adults, peripheral blood stem cells (PBSC) and bone marrow (BM) grafts, as well as mismatched and matched unrelated and matched related donors; all have involved the administration of four IV doses of abatacept, on days -1, +5, +14, and +28, in combination with standard calcineurin inhibitor-based GVHD prophylaxis. Collectively, the results to date suggest that this combination, including abatacept, very effectively prevents acute GVHD. However, these results also suggest that protection against chronic GVHD is more limited. In this current trial, the researchers will attempt to more effectively prevent chronic GVHD by extending the administration of abatacept, giving eight doses (additional doses days +56, +84, +112, and +150). This trial will test the hypothesis that extended abatacept administration (combined with a standard regimen of tacrolimus and mycophenolate mofetil) will effectively prevent acute and chronic GVHD in children and adolescents receiving URD HSCT, without compromising their engraftment or reconstitution of protective immunity to infection.

The ASCENT Trial is a single arm, multi-center, phase II study testing the hypothesis that extended abatacept administration (combined with a standard regimen of tacrolimus and mycophenolate mofetil) will effectively prevent acute and chronic GVHD in children and adolescents receiving URD HSCT, without compromising their engraftment or reconstitution of protective immunity to infection. The study will enroll 30 pediatric patients with serious NMHD undergoing URD HSCT. The trial will include two strata, based on donor matching. Stratum 1 will be for patients with 7/8 donors and stratum 2 will be for those with 8/8 (matched) donors. Study participants will be admitted to the hospital ten or eleven days prior to the day of transplant (day -10 or day -11) to complete a conditioning regimen to prevent the donor cells from being rejected. Patients will receive one of three reduced toxicity or intensity conditioning regimens based upon underlying disease and/or physician preference: (1) anti-thymocyte globulin, fludarabine, and a low dose of cyclophosphamide (FA patients only); (2) anti-thymocyte globulin, fludarabine, cyclophosphamide, and a low dose of total body radiation (SAA and other bone marrow failure disorders); or (3) alemtuzumab, fludarabine, melphalan, and thiotepa (hemoglobinopathy and non-SAA bone marrow failure disorders). All participants will receive 8 doses of abatacept (10 mg/kg intravenously on days -1, +5, +14, +28, +56, +84, +112, and +150). Recruitment is expected to last for about 2 years and participants will be followed for up to 3 years. Weight-based peripheral blood samples will be drawn longitudinally through two years to evaluate immune reconstitution.

The primary objective is to determine the rejection-free, severe graft-versus-host disease (GVHD)-free survival in pediatric patients with serious non-malignant hematologic diseases (NMHD) undergoing unrelated donor (URD) hematopoietic stem cell transplantation (HSCT) with abatacept added to conventional GVHD prophylaxis. The secondary objective is to characterize the impact of abatacept on infection and the reconstitution of protective immunity to infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sickle cell disease (stratum 1) must be between the ages of 3-20.99 years and patients with other diseases (stratum 2) between the ages of 0-20.99 years at the time of admission for transplant.
* Must have one of the following diseases:

  * Glanzmann thrombasthenia
  * Chronic granulomatous disease
  * Severe congenital neutropenia (with resistance to granulocyte colony-stimulating factor (GCSF) or chronic requirement of GCSF doses ≥10 mcg/kg)
  * Leukocyte adhesion deficiency
  * Shwachman-Diamond syndrome
  * Diamond-Blackfan Anemia (DBA; transfusion dependent, including steroid failure or inability to wean steroids)
  * Thalassemia major
  * FA
  * Dyskeratosis congenita
  * Chediak Higashi syndrome
  * Acquired (immune; non-inherited, non-congenital) SAA
  * Any genotypic form of SCD with severe disease, defined as one or more of the following criteria:

    * Previous clinical stroke, as evidenced by a neurological deficit lasting longer than 24 hours, which is accompanied by radiographic evidence of ischemic brain injury and cerebral vasculopathy.
    * Asymptomatic cerebrovascular disease, as evidenced by one the following:

      * Progressive silent cerebral infarction, as evidenced by serial MRI scans that demonstrate the development of a succession of lesions (at least two temporally discreet lesions, each measuring at least 3 mm in greatest dimension on the most recent scan) or the enlargement of a single lesion, initially measuring at least 3 mm. Lesions must be visible on T2-weighted MRI sequences.
      * Cerebral arteriopathy, as evidenced by abnormal TCD testing (confirmed elevated velocities in any single vessel of time-averaged mean of the maximum velocity (TAMMV) > 200 cm/sec for non-imaging TCD) or by significant vasculopathy on magnetic resonance angiograph (MRA; greater than 50% stenosis of > 2 arterial segments or complete occlusion of any single arterial segment).
    * Frequent (3 or more per year for preceding 2 years) painful vaso-occlusive episodes (defined as episode lasting 4 hours or more and requiring hospitalization or outpatient treatment with parenteral opioids). If patient is on hydroxyurea and its use has been associated with a decrease in the frequency of episodes, the frequency should be gauged from the 2 years prior to the start of this drug.
    * Recurrent (3 or more in lifetime) acute chest syndrome events which have necessitated erythrocyte transfusion therapy.
    * Any combination of 3 or more acute chest syndrome episodes and vaso-occlusive pain episodes (defined as above) yearly for 3 years. If patient is on hydroxurea and its use has been associated with a decrease in the frequency of episodes, the frequency should be gauged from the 3 years prior to the start of this drug.
  * Other inherited or congenital marrow failure syndromes complicated by SAA
  * Other inherited or congenital red blood cell disorders requiring monthly chronic transfusion therapy.
  * Congenital platelet disorders requiring frequent platelet transfusions (patient must have received at least 10 transfusions in the last 3 years).
  * Other inherited or congenital granulocyte disorders resulting in at least three inpatient hospitalizations in the past three years for infection.
* Must have an unrelated adult donor (marrow or PBSC) who is a 7 or 8/8 match
* All patients and/or their parents or legal guardians must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.
* Must have been evaluated and adequately counseled regarding treatment options by a pediatric hematologist.
* Negative serum pregnancy test for females of childbearing potential only. Pregnancy must be excluded before the start of treatment with study drugs and prevented thereafter by reliable contraceptive methods.

Exclusion Criteria:

* HLA matched related donor
* Pulmonary dysfunction defined as diffusing capacity of the lungs for carbon monoxide (DLCO; corrected for hemoglobin), forced expiratory volume in one second (FEV1), or forced vital capacity (FVC) < 40% of predicted. In a child unable to perform pulmonary function testing, a chronic need for supplemental oxygen will serve as the exclusionary criterion.
* Renal dysfunction defined as estimated glomerular filtration rate (GFR) of <60 ml/min/1.73m2.
* Severe cardiac dysfunction defined as shortening fraction < 25%.
* Bridging (portal to portal) fibrosis or cirrhosis of the liver
* Clinical stroke within 6 months of anticipated transplant
* Karnofsky or Lansky functional performance score < 50%
* HIV infection
* Uncontrolled viral, bacterial, fungal, or protozoal infection at the time of study enrollment.
* Patient with unspecified chronic toxicity serious enough to detrimentally affect the patient's capacity to tolerate HSCT.
* Patient or patient's guardian(s) unable to understand the nature and risks inherent in the HSCT process.
* History of non-compliance severe enough in the estimation of the treating team to preclude the patient from undergoing unrelated donor transplantation.
* Patient is pregnant or lactating.
* Patient with a 7/8 URD donor and HLA antibody testing (see below) demonstrating an antibody directed against a donor disparate HLA molecule.

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | Up to 3 years
  Event-free survival is a composite endpoint defined as rejection-free, severe GVHD-free survival. Events for this outcome include death, severe (grade II-IV) acute GVHD up to day 100, moderate to severe chronic GVHD up to 1 year, and/or graft rejection up to 1 year.

SECONDARY OUTCOMES:
Cytomegalovirus (CMV) Viremia | Up to Day 180
  The number of participants experiencing cytomegalovirus (CMV) viremia will be reported. CMV viremia will be defined as the occurrence of a positive polymerase chain reaction (PCR) test prior to Day 180.
CMV Invasive Disease | Up to 2 years
  The number of participants experiencing CMV invasive disease will be reported. CMV invasive disease will be defined in accordance with the Blood and Marrow Transplant Clinical Trials Network Manual of Procedures.
Post-transplant lymphoproliferative disease (PTLD) | Up to 2 years
  The number of participants experiencing post-transplant lymphoproliferative disease (PTLD) will be reported. PTLD will be defined in accordance with the World Health Organization's (WHO) Classification of Tumours of Haematopoietic and Lymphoid Tissues.
Regimen-Related Toxicity | Day 42 Post-transplant
  The number of participants experiencing regimen-related toxicity (RRT) will be reported. RRT will be scored according to the Bearman scale. Major RRT, defined as grade 4 (causing death) in any organ system or grade 3 for pulmonary, cardiac, renal, oral mucosal, neurologic, or hepatic, will be recorded.
Neutrophil Recovery | Up to Day 60
  The time to neutrophil recover, in days, will be reported. Neutrophil recovery will be defined as the first of 3 consecutive days following the nadir that the absolute neutrophil count is at least 500/microliter of blood.
Platelet Recovery | Up to Day 60
  The time to platelet recover, in days, will be reported. Platelet recovery will be defined as the first day that the platelet count is at least 50,000/microliter of blood, without a transfusion in the preceding 7 days.
Non-Engraftment | Day 28
  The number of participants experiencing non-engraftment will be reported. Non-engraftment will be defined as lack of neutrophil recovery, or neutrophil recovery with lack of myeloid donor chimerism.
Secondary Graft Failure | Up to 3 years
  The number of participants experiencing secondary graft failure will be reported. Secondary graft failure will be defined by initial engraftment but subsequent development of an absolute neutrophil count (ANC) < 500/μl for fourteen consecutive days.
Graft Loss | Up to 3 years
  The number of participants experiencing graft loss will be reported. Graft loss will be defined by initial engraftment (assessed by neutrophil recovery and donor chimerism) with the subsequent loss of donor myeloid chimerism (regardless whether persistent neutropenia develops).
Acute GVHD | Up to 1 year
  The number of participants experiencing acute GVHD (including all grades and stratified by grades) will be reported. Acute GVHD will be assessed according to the Blood and Marrow Transplant Clinical Trials Network Manual of Procedures.
Chronic GVHD | Up to 2 years
  The number of participants experiencing chronic GVHD (including overlap syndrome) will be reported. Chronic GVHD will be assessed according to the Blood and Marrow Transplant Clinical Trials Network Manual of Procedures.
Immune Suppression-Free Survival | Year 2
  The number of participants experiencing immune suppression-free survival will be reported. Immune suppression-free survival is measured as participant survival while off all systemic immunosuppressive agents.
Immune Suppression-Free/Disease-Free Survival | Year 2
  The number of participants experiencing immune suppression-free/disease-free survival will be reported. Immune suppression-free/disease-free survival will be defined as rejection-free survival off all systemic immunosuppressive agents.
Rejection-free survival | Up to 3 years
  The number of participants experiencing rejection-free survival will be reported. Rejection-free survival will be defined as survival without non-engraftment, secondary graft failure, or graft loss.
Overall survival | Up to 3 years
  The number of participants experiencing surviving at the end of the study follow up period will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: John Horan, MD, Principal Investigator — Emory University
Locations (9):
- United States (9):
  - Children's of Alabama, Birmingham, Alabama
  - Nemours/Alfred I. DuPont Hospital for Children, Wilmington, Delaware
  - Childrens Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Mississippi Medical Center, Children's Center for Cancer and Blood Disorders, Jackson, Mississippi
  - Hackensack Meridian Health, Hackensack, New Jersey
  - Oishei Children's Hospital, Buffalo, New York
  - Columbia University Irving Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No